CLINICAL TRIAL: NCT05949879
Title: Dose Response Effects of Pecan Consumption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Professor, Director of UGA Obesity Initiative, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROJECT00007288
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Dyslipidemias; Overweight and Obesity; Nutrition, Healthy
MeSH Terms: conditions — Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Four groups of 28-day parallel feeding trials with three groups receiving different amounts of pecans (low, mid, high) and one group serving as control (instructed to maintain their current habitual diet and avoid any nut consumption for the 28-day intervention).
Who Masked: Participant
Masking Description: Participants are blinded to which group they are in and what oil they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pecan LOW (Experimental): Participants are given pecans and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: Pecan LOW
- Pecan MID (Experimental): Participants are given pecans and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: Pecan MID
- Pecan HIGH (Experimental): Participants are given pecans and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: Pecan HIGH
- CONTROL (Experimental): Participants are asked to maintain their current habitual diet and avoid any tree nut/peanut consumption for the entire 28-day intervention period.
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: Pecan LOW — Participants are provided with a quantity of pecans that delivers 6% of the participant's estimated energy needs for 28 days.
  Arms: Pecan LOW
Other: Pecan MID — Participants are provided with a quantity of pecans that delivers 13% of the participant's estimated energy needs for 28 days.
  Arms: Pecan MID
Other: Pecan HIGH — Participants are provided with a quantity of pecans that delivers 20% of the participant's estimated energy needs for 28 days.
  Arms: Pecan HIGH
Other: CONTROL — Participants are asked to maintain their current habitual diet and to avoid any tree nut/peanut consumption for the entire 28-day intervention period.
  Arms: CONTROL

SUMMARY:
The bioactive compounds contained in tree nuts have been shown to beneficially affect cardiometabolic health outcomes. Pecans contain more total phenols, sterols, and flavonoids than any other tree nut. They also are a rich source of polyunsaturated fatty acids (PUFAs), fiber, vitamin A, vitamin E, folic acid, calcium, magnesium, phosphorus, potassium, and zinc. These bioactive components in pecans are likely the reason for the previously documented improvements in cardiometabolic health.

The specific aims of this study are to:

* Examine the effect of pecan consumption at doses of 6%, 13%, and 20% of total energy needs on fasting and postprandial blood lipids.
* Examine the effect of pecan consumption at doses of 6%, 13%, and 20% of total energy needs on plasma markers associated with overall health.
* Examine the effect of pecan consumption at doses of 6%, 13%, and 20% of total energy needs on subjective and physiologic postprandial measures of hunger and satiety.

Participants will be asked to:

* Consume pecans daily for 28 days or maintain their current habitual diet.
* Attend three short weekly visits for fasting blood craws, body measurements, and collect their next week's supply of study materials.
* Attend two longer (5 h) testing visits which include consuming a standard breakfast meal and having their blood drawn periodically before and after breakfast.

Researchers will compare pecan LOW, pecan MID, pecan HIGH, and the Control group to examine the physiologic effects of incorporating various dosages of pecans into one's diet.

DETAILED DESCRIPTION:
Cardiovascular disease risk factors, including higher BMIs and poor cholesterol profiles, are on the rise and contribute to the United States' growing disease burden. Research investigating the relationship between pecan nut consumption and cardiometabolic outcomes has shown that pecan nut consumption can significantly benefit fasting and postprandial blood lipids, reduce CVD risk factors, promote weight maintenance, improve subjective and psychological markers of physiological appetite, increase total antioxidant capacity, and increase energy expenditure and fat oxidation. However, the current literature on pecan consumption and health outcomes only encompasses physiological benefits coming from a dosage of ~45g/day and above, which is above the current dietary guidelines. This study will be the first dose-response study examining the minimalist effective dose and determining the most effective dosage of pecan consumption on metabolic and cardiovascular outcomes. If lower doses of pecans in the diet are found to improve fasting and postprandial lipid metabolism and markers of chronic disease risk, these study findings could lead to improvements in health.

This prospective clinical study is a single-blinded, randomized control trial in adults at increased risk for cardiovascular disease (poor cholesterol profiles or overweight/obesity). There are four diet interventions: pecan LOW (6% energy from pecans), pecan MID (13% energy from pecans), pecan HIGH (20% energy from pecans), and CON (instructed to maintain their current habitual diet and abstain from any tree nut/peanut consumption for the duration of the intervention). This study protocol consists of a 28-day diet intervention that will involve substituting pecans for commonly consumed snack or meal items every day for the entire 28-day intervention or maintaining a current/usual diet.

There are a total of six testing visits: a screening visit (V0), a pre-intervention visit (V1), short weekly visits (end of weeks 1, 2, and 3; V2-V4), and a post-intervention visit (V5).

At screening (V0), qualification is confirmed based on anthropometrics and fasting blood draw, which is analyzed for a cholesterol panel and blood glucose. Additionally, energy requirements are estimated at this visit for use in the diet intervention.

At V1, participants will have anthropometrics measured, including body composition, by DEXA. Next, a certified phlebotomist places an IV catheter and takes the fasting blood sample. Then the participant consumes a high-saturated-fat meal challenge, delivering 17% of their estimated energy needs (from V0). Then the participant has blood drawn 7 times using the IV catheter over the next 4 hours.

The 28-day diet intervention will consist of research personnel providing pecans that deliver 6%, 13%, or 20% of the participant's daily energy needs (determined at V0). Participants placed in one of the three pecan diets will receive counseling at the baseline (V1) and weekly intervention visits (V2-V4) on substituting pecans for isocaloric foods from their habitual diet. Individuals randomized in the control group will be instructed to follow their habitual diet and will not be provided with any food items.

Participants return weekly (V2, V3, V4) to return study materials and collect food for the next week (if applicable). At these weekly visits, participants also have a fasting blood draw, and researchers will collect the participant's body measurements.

At the end of the 28-day dietary intervention, participants return for V5, where all procedures from V1 are repeated.

The investigators hypothesize that diets including the daily consumption of pecans will benefit health outcomes and lower cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 75-year-old men and women at increased risk of cardiovascular disease. Increased risk of cardiovascular disease will be defined by either elevated cholesterol profiles or overweight/obesity.
* Elevated cholesterol profiles will be defined as: "Borderline High" and/or "at risk" in two or more of the following variables (total cholesterol: 180-239 mg/dL, LDL cholesterol 110- 159 mg/dL, triglycerides 130-199 mg/dL) --or---"High" in total cholesterol (240 mg/dL and higher), LDL (160 mg/dL or higher), or triglycerides (between 200-350 mg/dl).
* Overweight/obesity will be defined by body mass index (overweight > 28 kg/m2 or obesity 30 kg/m2 or greater).

Exclusion Criteria:

* Probable familial hypercholesterolemia, defined by: total cholesterol greater than 290 mg/dL or LDL levels greater than 190 mg/dL plus a family history of myocardial infarction (MI) before 50 years of age in a 2nd-degree relative or below age 60 in a 1st-degree relative
* Alcohol intake >3 drinks/d for males or >2 drinks/d for females
* Individuals with food allergies/sensitivities to foods provided in the study, including tree nuts, gluten, and or lactose/dairy
* Individuals who regularly consume nuts and/or nut butter (defined as consumption of >2 servings (~56g) of tree nuts, nuts, or nut butter (e.g., peanut butter, almond butter) per week
* Individuals adhering to special diets, including, but not limited to, the ketogenic diet, intermittent fasting, vegetarian diet, or carbohydrate-restricted diets
* Plans to begin a weight loss/exercise regime during the trial
* Weight gain or loss of more than 5% of their body weight in the past 3 months
* History of previous or current renal or bowel disease
* Females who are currently pregnant or lactating
* Individuals participating in >3 hours/week of exercise
* Women on hormone replacement therapy for <2 years
* Fasting glucose >126 mg/dL
* Blood pressure >180/120 mmHg
* History of medical or surgical events that could affect digestion or swallowing
* Gastrointestinal surgery, atherosclerosis, or bleeding disorders
* Tobacco or nicotine use
* Previous heart attack (MI) or stroke, previous or current diagnosis of cancer
* Chronic or metabolic diseases
* Medication use affecting digestion and absorption, medications affecting metabolism (e.g., thyroid meds), lipid-lowering medications, medications for diabetes, blood thinning medications
* Steroid/hormone therapies or current antibiotic cycles

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in fasting serum lipoprotein and cholesterol concentrations | Baseline, 4 weeks
  The concentration of fasting serum total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and apolipoprotein B (mg/dl).
Change in fasting serum lipoprotein particle numbers | Baseline, 4 weeks
  The number of particles of low-density lipoproteins (LDL), LDL small, HDL large, LDL medium, lipoprotein (a) (nmol/L).
Change in fasting and postprandial plasma triglyceride concentrations | Baseline, 4 weeks
  The concentration of plasma triglycerides before and after the high saturated fat meal challenge at both pre-and post-intervention visits (mg/dL).
Change in fasting and postprandial plasma non-esterified fatty acid (NEFA) concentrations | Baseline, 4 weeks
  The concentration of plasma NEFAs before and after the high saturated fat meal challenge at both pre-and post-intervention visits (mEq/L).
Change in fasting and postprandial plasma glucose concentrations | Baseline, 4 weeks
  The concentration of plasma glucose before and after the high saturated fat meal challenge at both pre-and post-intervention visits (mg/dL).
Change in fasting and postprandial plasma insulin concentrations | Baseline, 4 weeks
  The concentration of plasma insulin before and after the high saturated fat meal challenge at both pre-and post-intervention visits (uU/mL).
Change in fasting and postprandial plasma appetite control hormones concentrations | Baseline, 4 weeks
  The concentration of plasma appetite control hormones before and after the high saturated fat meal challenge at both pre-and post-intervention visits. Appetite control hormones include Cholecystokinin (CCK), Peptide YY (PYY), and Ghrelin (pg/mL).
Change in fasting and postprandial subjective feelings related to appetite | Baseline, 4 weeks
  Visual analog scale ratings of feelings related to appetite before and after the high saturated fat meal challenge at both pre-and post-intervention visits. Subjective feelings of hunger, fullness, desire to eat, prospective consumption, and a composite appetite score are measured by visual analog scales (mm).
Change in fasting and postprandial plasma Malondialdehyde (MDA) | Baseline, 4 weeks
  The concentration of MDA before and after the high saturated fat meal challenge at both pre-and post-intervention visits (nmol/mL).
Change in fasting and postprandial plasma total antioxidant capacity | Baseline, 4 weeks
  Total antioxidant capacity before and after the high saturated fat meal challenge at both pre-and post-intervention visits (U/mL).
Change in fasting and postprandial plasma antioxidant parameters | Baseline, 4 weeks
  Glutathione peroxidase activity, superoxide dismutase activity, and glutathione-s-transferase activity before and after the high saturated fat meal challenge at both pre-and post-intervention visits (U/mL).
Change in fasting and postprandial plasma inflammatory cytokine concentrations | Baseline, 4 weeks
  The concentration of interleukin-1 beta, C reactive protein, tumor necrosis factor-alpha, and interleukin-6 before and after the high saturated fat meal challenge at both pre-and post-intervention visits (pg/mL).
Change in fasting and postprandial plasma markers of coagulation potential | Baseline, 4 weeks
  The concentration of plasminogen activator inhibitor-1 and tissue factor before and after the high saturated fat meal challenge at both pre-and post-intervention visits (pg/mL).
Change in fasting and postprandial plasma angiopoietin-like (ANGPTL) proteins | Baseline, 4 weeks
  The concentration of ANGPTL 3, ANGPTL 4, and ANGPTL 8 before and after the high saturated fat meal challenge at both pre-and post-intervention visits (ng/mL).
Change in fasting insulin resistance metrics | Baseline, 4 weeks
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) and Homeostatic Model Assessment for β-cell function (HOMA-B) will be calculated from fasting insulin and glucose measures before and after the 28-day intervention.

SECONDARY OUTCOMES:
Change in fasting serum hepatic enzymes | Baseline, 4 weeks
  Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), and Gamma-Glutamyl Transferase (GGT) (U/L).
Change in fasting serum hepatic proteins | Baseline, 4 weeks
  Total protein and albumin (g/dL).
Change in fasting serum bilirubin | Baseline, 4 weeks
  Total total bilirubin, direct bilirubin, and indirect bilirubin (mg/dL).
Change in additional fasting and postprandial plasma inflammatory cytokine concentrations | Baseline, 4 weeks
  The concentration of monocyte chemoattractant protein-1 and interleukin-10 before and after the high saturated fat meal challenge at both pre-and post-intervention visits (pg/mL).
Change in additional fasting and postprandial plasma markers of coagulation potential | Baseline, 4 weeks
  The concentration of Von Willebrand factor, tissue factor pathway inhibitor, fibrinogen, and D-dimer before and after the high saturated fat meal challenge at both pre-and post-intervention visits (pg/mL).
Change in overall liking and desire to consume subjective ratings of the intervention food provided | Baseline, Week 1, Week 2, Week 3, Week 4
  Visual analog scale ratings of feelings related to overall liking and desire to consume the intervention food are measured by visual analog scales (mm).
Change in acute dietary intake | Baseline, 4 weeks
  One-day food logs will be used to record all foods and beverages consumed on testing days.

OTHER OUTCOMES:
Change in blood pressure | Baseline, 4 weeks
  Systolic and diastolic blood pressure (mmHg).
Change in body weight | Baseline, 4 weeks
  Body weight (kg).
Change in body composition | Baseline, 4 weeks
  DEXA will be used to measure body fat percentage (body fat %).
Change in diet composition | Baseline, Week 2, Week 4
  3-day food logs will be used to record foods and beverages consumed before and during the 28-day intervention period.
Change in fasting and postprandial fatty acid composition | Baseline, 4 weeks
  Fatty acid composition of plasma before and after the high saturated fat meal challenge at pre- and post-intervention visits (% total triglycerides).
Change in fasting tocopherol concentrations | Baseline, 4 weeks
  Plasma tocopherol concentrations (ug/ml).
Change in fasting urolithin concentrations | Baseline, 4 weeks
  Plasma urolithin concentrations (ng/mL).
Change in anthropometric circumferences | Baseline, 4 weeks
  Hip and waist circumferences (cm).
Change in resting metabolic rate | Screening
  Resting metabolic rate (RMR) will be measured for 30 minutes on the TrueOne 2400 (Parvo Medics, Sandy, UT).
Change in perceived stress | Baseline, 4 weeks
  A Perceived Stress Scale (PSS) will be administered and scored to determine stress levels.
Change in anxiety | Baseline, 4 weeks
  The State-Trait Anxiety Inventory (STAI) will be administered and scored to determine anxiety levels.
Change in self-reported physical activity levels | Baseline, Week 2, Week 4
  The International Physical Activity Questionnaire will be used to collect self-reported average physical activity levels (met/min).
Change in self-reported consumption of the intervention food or foods similar to the intervention food | Baseline, 4 weeks
  A 4-week post questionnaire will be used to collect self-reported intake of the intervention food or foods similar to the intervention food.
Change in body Mass Index (BMI) | Baseline, 4 weeks
  BMI will be calculated based on height and weight measures (kg/m2).
Change in self-reported dietary intake | Screening
  The Diet History Questionnaire III (DHQ III) is an NIH food frequency questionnaire that consists of 135 food and beverage line items and 26 dietary supplement questions. The DHQ III will be used to assess food and dietary supplement intakes prior to participation in the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie A Cooper, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

REFERENCES:
- [Derived] Guadagni AJ, Paton CM, Cooper JA. Dose Response Effects of Pecan Consumption on Blood Lipid Profiles in Adults with Excess Body Weight and/or Dyslipidemia: A Randomized Controlled Trial. J Nutr. 2026 Feb 4:101396. doi: 10.1016/j.tjnut.2026.101396. Online ahead of print. PMID 41651071